CLINICAL TRIAL: NCT01100424
Title: Assessment of Tear Film-Based Proteins Associated With Care Solution Induced Corneal Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMA-09-20
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-07

CONDITIONS: Corneal Staining
Keywords: Contact lenses; Contact lens solution; Corneal staining

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact lens wearers (Experimental): Contact lens wearers experienced three currently available contact lens/contact lens care combinations in randomized order: balafilcon A + Optifree RepleniSH, balafilcon A + ReNu MultiPlus, and balafilcon A + Unisol 4 saline.
  Interventions: Device: Opti-Free RepleniSH; Device: ReNu MultiPlus; Device: Balafilcon A; Other: Unisol 4
- Non-lens wearers (No Intervention): Non-lens wearers completed one study visit and served as the control group.

INTERVENTIONS:
Device: Opti-Free RepleniSH — Commercially available contact lens solution used for pre-soaking balafilcon A contact lenses overnight prior to lens insertion.
  Arms: Contact lens wearers
Device: ReNu MultiPlus — Commercially available contact lens solution used for pre-soaking balafilcon A contact lenses overnight prior to lens insertion.
  Other Names: Renu
  Arms: Contact lens wearers
Device: Balafilcon A — Commercially available silicone hydrogel contact lenses removed from blister pack and soaked overnight in Opti-Free Replenish, ReNu MultiPlus, or Unisol 4, then applied to the eye and worn for 2 hours.
  Other Names: PureVision
  Arms: Contact lens wearers
Other: Unisol 4 — Commercially available non preserved sterile saline solution used for pre-soaking balafilcon A contact lenses overnight prior to lens insertion.
  Arms: Contact lens wearers

SUMMARY:
The purpose of this study was to investigate the association of inflammatory mediators found in the tear film during the development and following the induction of contact lens solution-induced corneal staining.

ELIGIBILITY:
Inclusion Criteria:

For non-lens wearers:

* Normal eyes.
* Currently not wearing contact lenses and has not worn contact lenses for the previous 6 months.
* Free of dry eye using the Ocular Surface Disease Index (Schiffman et al).
* Other protocol-defined inclusion criteria may apply.

For contact lens wearers:

* Currently wearing soft contact lenses.
* Free of dry eye during lens wear using the Contact Lens Dry Eye Questionnaire Short-Form (Nichols et al, Cornea, 2002).
* Reports a contact lens wearing time of at least 12 hours per day, 7 days per week, daily wear basis (not overnight wear).
* Reports only occasional use of contact lens rewetting drops or artificial tears.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

For non-lens wearers and contact lens wearers:

* Pregnant.
* Participating in another research study.
* Exhibiting staining with fluorescein in more than 5% of the total cornea (graded by "extent" of staining across 5 regions).
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Tear Protein Expression | 1 day

SECONDARY OUTCOMES:
Corneal Staining | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, Study Director — Alcon, Ltd.
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States